CLINICAL TRIAL: NCT00366288
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PAZ-417 Administered Orally to Healthy Young and Healthy Elderly Subjects
Brief Title: Study Evaluating PAZ-417 in Healthy Young/Elderly
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 3186A1-100
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Alzheimer Disease
Keywords: Healthy; Safety
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — plasma and urine

GROUPS / COHORTS (7):
- 1
  Interventions: Drug: PAZ-417
- 2
  Interventions: Drug: PAZ-417
- 3
  Interventions: Drug: PAZ-417
- 4
  Interventions: Drug: PAZ-417
- 5
  Interventions: Drug: PAZ-417
- 6
  Interventions: Drug: PAZ-417
- 7
  Interventions: Drug: PAZ-417

INTERVENTIONS:
Drug: PAZ-417 — 2.5 mg, 5, 10, 25, 50 mg - fasted in healthy young 10 mg - food effect in healthy young 5 and 25 mg -fasted healthy elderly.

SUMMARY:
This study is to evaluate the safety and tolerability of single, ascending doses of PAZ-417 in healthy young and healthy elderly subjects. The effect of a high fat meal on the metabolism of PAZ-417 will also be studied, along with blood levels of PAZ-417 . Changes in cognitive function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, aged 18 to 50 years inclusive (healthy young subjects) and > 65 years inclusive (elderly subjects) on study day 1. Women of nonchildbearing potential may be included if they are either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for ≥1 year (with estradiol ≤25 pg/mL[92 pmol/L] and FSH ≥40 mIU/mL) and must have a negative serum pregnancy test result within 48 hours before administration of test article. Women who are surgically sterile or post-menopausal must provide documentation of the procedure by an operative report or by ultrasound and have a negative serum pregnancy test result within 48 hours before administration of test article.
2. The elderly subjects must be generally healthy, but may be enrolled with a stable, chronic illness, if it is well-controlled, and does not interfere with the primary objective of the study. Subjects may be included with clinically important deviations from normal limits in medical history, physical examination, vital signs, 12-lead ECGs, or clinical laboratory test results which are associated with stable, chronic, well-controlled, medical conditions.
3. The estimated creatinine clearance must be within the age-appropriate normal range.

Exclusions Criteria:

1. Presence or history of any disorder that may prevent the successful completion of the study.
2. Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article.
3. Exclude subjects with a history of vascular disorders (peripheral, coronary, venous), chronic inflammatory disorders (e.g., rheumatoid arthritis), hematologic disorders, and bleeding disorders (e.g., hemophilia, idiopathic thrombocytopenic purpura, von willebrand's disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of a certain town
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Phoenix, Arizona, United States